CLINICAL TRIAL: NCT07009808
Title: Effects of Different Doses of Nalbuphine on Anxiety and Depression in Patients Undergoing Ectopic Pregnancy Surgery: A Prospective, Randomized, Controlled Study
Brief Title: Nalbuphine Dosing and Its Impact on Anxiety and Depression in Ectopic Pregnancy Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu Jinjiang Maternity and Child Health Hospital (Other)
Responsible Party: Principal Investigator, Fei Jia, Director of Anesthesiology Department, Chengdu Jinjiang Maternity and Child Health Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202427
Record Dates: First submitted 2025-05-27; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Ectopic Pregnancy; Anxiety; Depression; Nalbuphine
Keywords: Ectopic Pregnancy; Anxiety; Depression; Nalbuphine
MeSH Terms: conditions — Pregnancy, Ectopic; Anxiety Disorders; Depression | interventions — Nalbuphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study employs a randomized, double-blind design to ensure that both the participants and the assessors are unaware of their respective treatment assignments. All patients will be randomly assigned to three groups, receiving different concentrations of nalbuphine via a pain management pump, while the researchers conducting postoperative evaluations (including anxiety, depression, and pain scores) will remain blind to the specific group assignments. Data analysis will also be conducted in a blinded manner to minimize bias. This comprehensive masking approach aims to ensure the objectivity and reliability of the study's results, accurately assessing the impact of nalbuphine on postoperative psychological and pain management in patients with ectopic pregnancy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- N1 Group (Experimental): Patients in this group will receive Nalbuphine at a concentration of 0.20 mg/ml, totaling 30 mg, combined with 10 mg of Metoclopramide for postoperative analgesia. This group aims to evaluate the effects of this specific dosing on anxiety and depression levels following ectopic pregnancy surgery.
  Interventions: Drug: Nalbuphine 0.20mg/ml(total 30 mg)
- N2 Group (Experimental): articipants in this group will be administered Nalbuphine at a concentration of 0.27 mg/ml, totaling 40 mg, along with 10 mg of Metoclopramide for postoperative pain management. The focus will be on assessing the impact of this dosage on the patients' anxiety and depression scores post-surgery.
  Interventions: Drug: Nalbuphine 0.27mg/ml(total 40 mg)
- N3 Group (Experimental): Individuals in this group will receive Nalbuphine at a concentration of 0.33 mg/ml for a total of 50 mg, paired with 10 mg of Metoclopramide for effective postoperative analgesia. This group will help determine the effects of this higher dosage on levels of anxiety and depression after surgery for ectopic pregnancy.
  Interventions: Drug: Nalbuphine 0.33mg/ml(total 50 mg)

INTERVENTIONS:
Drug: Nalbuphine 0.20mg/ml(total 30 mg) — In this group, participants will receive an intravenous infusion of Nalbuphine at a concentration of 0.20 mg/ml, which delivers a total of 30 mg over the course of 48 hours. Additionally, 10 mg of Metoclopramide will be administered to manage potential postoperative nausea. This intervention aims to assess the analgesic efficacy and its subsequent effect on psychological outcomes, specifically anxiety and depression, in patients undergoing surgery for ectopic pregnancy.
  Arms: N1 Group
Drug: Nalbuphine 0.27mg/ml(total 40 mg) — Participants assigned to this group will be treated with an intravenous infusion of Nalbuphine at a concentration of 0.27 mg/ml, resulting in a total dosage of 40 mg administered during the 48-hour postoperative period. They will also receive 10 mg of Metoclopramide to mitigate nausea and vomiting. This intervention is designed to evaluate the effectiveness of this dose in pain management and its influence on anxiety and depression levels post-surgery.
  Arms: N2 Group
Drug: Nalbuphine 0.33mg/ml(total 50 mg) — In this group, subjects will receive Nalbuphine at a concentration of 0.33 mg/ml, totaling 50 mg, delivered through intravenous infusion for 48 hours. Along with this, 10 mg of Metoclopramide will be included to address potential postoperative discomfort. This intervention seeks to explore how this higher concentration impacts pain relief and subsequent psychological effects, specifically targeting anxiety and depression following ectopic pregnancy surgery.
  Arms: N3 Group

SUMMARY:
This prospective, randomized, controlled study aims to evaluate the impact of different doses of nalbuphine on anxiety and depression in patients undergoing surgery for ectopic pregnancy. Ectopic pregnancy, which occurs in approximately 2% of all pregnancies, often requires surgical intervention, leading to potential psychological distress such as anxiety and depression in affected women. Effective postoperative pain management is essential to enhance recovery and reduce emotional disturbances.

The study will involve 165 eligible patients diagnosed with ectopic pregnancy at Jinjiang District Maternal and Child Health Hospital. Participants will be randomly assigned to three groups, each receiving a different concentration of nalbuphine combined with metoclopramide for postoperative analgesia. The primary outcome will focus on changes in anxiety and depression scores measured on postoperative day three, while secondary outcomes will assess pain levels, the use of patient-controlled analgesia (PCA), the necessity for rescue analgesics, and the occurrence of adverse reactions.

Sample size calculations suggest that at least 165 participants are required to achieve adequate statistical power. Data will be analyzed using SPSS 25.0 software, with results expected to provide insights into the effectiveness of nalbuphine in improving postoperative recovery and mental health in women experiencing ectopic pregnancy. The study has received ethical approval and is funded by the Chengdu Medical Research Projects (No. 2023465, 2022548, and 2023304).

DETAILED DESCRIPTION:
Background:

Ectopic pregnancy occurs when a fertilized egg implants outside the uterine cavity, affecting approximately 2% of all pregnancies. Surgical intervention is the primary treatment, which can lead to significant psychological effects, including anxiety and depression. Studies indicate that patients may experience various emotional disturbances post-surgery, negatively impacting their social adaptability and interpersonal relationships. Effective postoperative pain management is crucial for recovery and may also help alleviate these emotional challenges. Nalbuphine, an opioid receptor agonist-antagonist that primarily acts on the kappa receptor, has been shown to provide pain relief with a lower incidence of respiratory depression and may have a positive impact on mental health compared to traditional opioids.

Objective:

The main objective is to investigate the effects of different concentrations of nalbuphine on anxiety and depression in patients with ectopic pregnancy post-surgery, focusing on changes in anxiety and depression scores on postoperative day three. The secondary objective is to compare the postoperative analgesic effects and the incidence of adverse reactions associated with different concentrations of nalbuphine.

Methods:

This study is designed as a single-center, prospective, randomized, controlled clinical trial conducted at Jinjiang District Maternal and Child Health Hospital. Ethical approval will be obtained, and all participants will provide informed consent.

Interventions:

165 eligible patients will be randomly assigned into three groups (N1, N2, N3), each receiving different doses of nalbuphine combined with metoclopramide for postoperative pain management, with a total volume of 150ml for each group. The groups are as follows:

* Group A: Nalbuphine 0.20 mg/ml (total 30 mg)
* Group B: Nalbuphine 0.27 mg/ml (total 40 mg)
* Group C: Nalbuphine 0.33 mg/ml (total 50 mg)

Patient-controlled analgesia (PCA) will be maintained for 48 hours.

Primary Outcome:

The primary outcome will be the assessment of anxiety and depression scores measured on postoperative day three.

Secondary Outcomes:

Secondary outcomes will include:

1. Visual Analog Scale (VAS) resting and activity pain scores at multiple time points (T1: 6 hours, T2: 12 hours, T3: 24 hours, T4: 48 hours).
2. Number of PCA button presses.
3. Use and frequency of rescue analgesics.
4. Incidence of adverse reactions such as drowsiness, dizziness, nausea, vomiting, and respiratory depression.
5. Time to mobilization and time to first flatus.

Ethics Approval:

This study has received approval from the ethics committee of Chengdu Jinjiang District Maternal and Child Health Hospital (Approval Number: 202312). All participants must sign an informed consent form to ensure the respect of participant rights and data confidentiality. The study will strictly adhere to relevant ethical standards and legal regulations to protect participant safety and privacy.

Funding:

The study is funded by the Chengdu Medical Research Projects (No. 2023465, 2022548, and 2023304).

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of ectopic pregnancy, aged ≥18 years, and with normal psychological status.
2. Patients planned to undergo single-port laparoscopic surgery under general anesthesia, followed by postoperative patient-controlled intravenous analgesia (PCIA).
3. Patients classified as ASA I or II.
4. Able to understand the study process and methods, voluntarily participate, and sign the informed consent form.

Exclusion Criteria:

1. Patients using other analgesic methods or multiple analgesic approaches.
2. Patients with a history of allergies or allergies to anesthetic drugs.
3. Patients with a history of depression or mental illness.
4. Patients with other severe organ dysfunction.
5. Patients unable to operate the intravenous analgesia pump independently.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is exclusively for female participants, as ectopic pregnancy is a condition that occurs only in women.
Enrollment: 165 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2025-10-22 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative Anxiety and Depression Scores | Day 3 post-surgery
  The primary outcome of this study is to evaluate the levels of anxiety and depression in patients following surgery for ectopic pregnancy. This will be assessed using the Hospital Anxiety and Depression Scale (HADS) at the following specific time point:

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) Pain Scores | Postoperative 6 hours, 12 hours, 24 hours, and 48 hours
  This study will utilize the Visual Analog Scale (VAS) to assess pain levels in patients both at rest and during activity. Pain scores will be measured at the following specific time points to evaluate the efficacy of different dosages of nalbuphine in managing postoperative pain:
  T1: 6 hours post-surgery T2: 12 hours post-surgery T3: 24 hours post-surgery T4: 48 hours post-surgery
Effective Presses of the Pain Pump | 48 hours post-surgery
  The number of effective presses of the pain pump will be recorded for each patient during their hospital stay to evaluate the effectiveness of the pain pump in alleviating postoperative pain.
Need for Rescue Analgesia | 48 hours post-surgery
  This outcome will document whether patients require additional rescue analgesia postoperatively to assess the adequacy of the initial analgesic regimen.
Number of participants experience feelings of drowsiness | day 2 post-surgery
  Patients may feel unusually tired or sleepy after surgery. This can affect their attention and reaction times, increasing the risk of falls or other accidents.
Time to Ambulate | Perioperative
  This outcome will measure the time taken for patients to ambulate (get out of bed)
Time to Flatus | Perioperative
  This outcome will measure the time taken to pass gas post-surgery.
Number of participants experience feelings of Dizziness | day 2 post-surgery
  Patients might experience feelings of dizziness or loss of balance. This reaction can lead to discomfort and potential dangers when the patient is standing or walking.
Number of participants experience feelings of Nausea | day 2 post-surgery
  Patients may experience a sensation of wanting to vomit or feelings of nausea. This can impact their appetite and contribute to further discomfort.
Number of participants experience feelings of Vomiting | day 2 post-surgery
  In some cases, nausea may develop into vomiting, leading patients to actually expel contents from their stomach. This can affect recovery and may lead to dehydration or electrolyte imbalances.

IPD SHARING:
Plan to Share IPD: No
For our study "Effects of Different Doses of Nalbuphine on Anxiety and Depression in Patients Undergoing Ectopic Pregnancy Surgery: A Prospective, Randomized, Controlled Study" we have decided not to share Individual Participant Data (IPD). This decision is due to privacy concerns, data security requirements, ethical approval limitations, legal restrictions, and the study's design which did not accommodate data sharing. We believe this aligns with ethical standards and operational capabilities.

REFERENCES:
- [Background] Bollig KJ, Friedlander H, Schust DJ. Ectopic Pregnancy and Lifesaving Care. JAMA. 2023 Jun 20;329(23):2086-2087. doi: 10.1001/jama.2023.7292. PMID 37261808
- [Background] Farren J, Jalmbrant M, Falconieri N, Mitchell-Jones N, Bobdiwala S, Al-Memar M, Tapp S, Van Calster B, Wynants L, Timmerman D, Bourne T. Posttraumatic stress, anxiety and depression following miscarriage and ectopic pregnancy: a multicenter, prospective, cohort study. Am J Obstet Gynecol. 2020 Apr;222(4):367.e1-367.e22. doi: 10.1016/j.ajog.2019.10.102. Epub 2019 Dec 13. PMID 31953115
- [Background] Farren J, Jalmbrant M, Falconieri N, Mitchell-Jones N, Bobdiwala S, Al-Memar M, Tapp S, Van Calster B, Wynants L, Timmerman D, Bourne T. Differences in post-traumatic stress, anxiety and depression following miscarriage or ectopic pregnancy between women and their partners: multicenter prospective cohort study. Ultrasound Obstet Gynecol. 2021 Jan;57(1):141-148. doi: 10.1002/uog.23147. PMID 33032364
- [Background] Pan X, Wang J, Lin Z, Dai W, Shi Z. Depression and Anxiety Are Risk Factors for Postoperative Pain-Related Symptoms and Complications in Patients Undergoing Primary Total Knee Arthroplasty in the United States. J Arthroplasty. 2019 Oct;34(10):2337-2346. doi: 10.1016/j.arth.2019.05.035. Epub 2019 May 28. PMID 31229373
- [Background] Akshat S, Ramachandran R, Rewari V, Chandralekha, Trikha A, Sinha R. Morphine versus Nalbuphine for Open Gynaecological Surgery: A Randomized Controlled Double Blinded Trial. Pain Res Treat. 2014;2014:727952. doi: 10.1155/2014/727952. Epub 2014 Apr 14. PMID 24834352
- See also: Related Info — https://ccj.pku.edu.cn/article/info?aid=209401918
- See also: Related Info — https://www.jjfck.com/